CLINICAL TRIAL: NCT01178957
Title: Very-Low-Density-Lipoprotein-Triglyceride(VLDL-TG) Metabolism During Acute Hyperglycemia
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: ES-0004
Record Dates: First submitted 2010-04-21; First posted 2010-08-10 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Very-Low-Density-Lipoprotein(VLDL); Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Type 1 diabetes
  Interventions: Other: Hyperglycemia

INTERVENTIONS:
Other: Hyperglycemia — Hyperglycemia with a blood glucose of 15 mmol/L

SUMMARY:
The purpose of this study is to estimate the acute effect of hyperglycemia on Very-Low-Density-Lipoprotein-triglyceride(VLDL-TG) secretion.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes
2. Age 18-50 years

Exclusion Criteria:

1. Smoking
2. Alcohol abuse
3. Use of medications (except insulin in diabetics)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Type 1 diabetics
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Very-Low-Density-Lipoprotein-Triglyceride(VLDL-TG) secretion | 8 hours
  Very-Low-Density-Lipoprotein-Triglyceride(VLDL-TG) kinetics over a single study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology MEA, Aarhus Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Johansen RF, Sondergaard E, Sorensen LP, Nellemann B, Christiansen JS, Nielsen S. Isolated hyperglycaemia does not increase VLDL-triacylglycerol secretion in type 1 diabetic men. Diabetologia. 2015 Feb;58(2):355-62. doi: 10.1007/s00125-014-3422-6. Epub 2014 Nov 11. PMID 25385409